CLINICAL TRIAL: NCT00313469
Title: Sources of the Variability of the Response to Fluindione in Elderly Patients (PREPA) [Etude Des Sources de variabilité de la réponse à la Fluindione Chez Les Personnes âgées de 80 Ans et Plus (PREPA) ]
Brief Title: Sources of the Variability of the Response to Fluindione in Elderly Patients (PREPA)
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); GIS Institut de la Longévité (Unknown)
Responsible Party: Principal Investigator, France Mentré, Professor, Assistance Publique - Hôpitaux de Paris
Other Study IDs: INSERM; GIS Institut Longévité 2003
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Cardiovascular Disease
Keywords: Pharmacokinetics/Pharmacodynamics; Elderly; Anticoagulants
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for the measure of drug concentrations Blood samples with DNA measurements
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We propose to study the pharmacokinetic (PK) and pharmacodynamic (PD) components of the response to fluindione, the main oral anticoagulant used in France, in patients over 80.

We expect to gain a better understanding of the role of age, nutritional status, genetic factors and drug interactions in the variability of the response to fluindione.

DETAILED DESCRIPTION:
Oral anticoagulant drugs have improved the prognosis of patients with thromboembolic disease. However, optimal oral anticoagulation control is usually hampered by significant interindividual variability coupled with a narrow therapeutic window. In the elderly, this variability is enhanced by concurrent medications, nutritional status and physical condition. Age itself correlates with increased severity of complications, and adverse events due to anticoagulant drug are thought to be responsible for up to 5000 deaths a year in France.

Although half the patients receiving anticoagulant treatment are over 80, there has been only one study targeting this population so far. We therefore propose to study the pharmacokinetic (PK) and pharmacodynamic (PD) components of the response to fluindione, the main oral anticoagulant used in France, in patients over 80.

150 patients beginning fluindione treatment (or resuming after 2 weeks rest) will be recruited in the following departments: Geriatric, Cardiology, Nephrology, Cardiac Surgery, Internal Medicine (CHU Bichat-Claude Bernard, Paris) and Metabolic Diseases and Internal Medicine (CHU d'Angers). Blood sampling will take place before the beginning of the study (J0) to measure baseline INR and coagulation factors II and VII. Fluindione concentrations will also be measured in non-naive patients. INR, coagulation factors and fluindione will be measured at J2, J4, J6, J8, and twice weekly until they leave the hospital or up to a month. Many covariates will be recorded: age, gender, concurrent medications, biochemical analyses, functional and nutritional status. We will also investigate genetic factors by collecting DNA to genotype polymorphisms related to the target of the drug. Recent work has shown that both the response to common anticoagulant drugs and their metabolism was influenced by genetic polymorphisms, and there is now convincing evidence that drug targets are controlled by genetic polymorphisms which can play a major role in the variability of the response.

Throughout the study, the physicians remain free to adapt drug regimen and prescribe additional INR measurements.

Data analysis will be performed in INSERM Unit 738 (CHU Bichat-Claude Bernard) using nonlinear mixed-effect models, statistical techniques allowing the analysis of sparse data while quantifying the sources of variability.

We expect to gain a better understanding of the role of age, nutritional status, genetic factors and drug interactions in the variability of the response to fluindione. We will also assess whether measuring the activity of coagulation factors helps to anticipate dangerous increases in INR. These goals are vital to provide better care of the elderly and minimise costs arising from the frequency of severe side-effects.

Future perspectives include the development of a software and recommendations to help adapt anticoagulant treatment in the elderly, taking into account their condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients over and including 80 years old
* Hospitalised in one of the recruiting centers
* Initiating a treatment with fluindione (either first time or after more than 15 days holidays)

Exclusion Criteria:

* Contraindication to fluindione or one of its components
* Patients receiving other medications known to interfere with fluindione and preventing its use
* Patients with physical or mental impairment preventing them from signing the consent form
* Patients whose length of stay in hospital is less than 3 days

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people (>80 years) initiating a treatment with fluindione
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: France Mentré, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - CHU d'Angers, Angers
  - Hôpital Bichat-Claude Bernard, Paris